CLINICAL TRIAL: NCT04129866
Title: Mobile Interpretation Bias Modification Clinical Trial
Acronym: M-IBM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Southern Mississippi (Other)
Collaborators: Military Suicide Research Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH-16-2-0004
Record Dates: First submitted 2019-10-10; First posted 2019-10-17 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Anxiety Sensitivity; Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M-IBM (Experimental): M-IBM is based on a slightly modified version of the word sentence association paradigm focused on words and sentences related to common concerns among those with elevated anxiety sensitivity cognitive concerns (i.e., losing control of mental processes).
  Interventions: Behavioral: M-IBM
- Control IBM (Placebo Comparator): Control-IBM is identical to M-IBM except that the sentence that follows the cue word is not related to an anxious-threat interpretation of the cue word.
  Interventions: Behavioral: Control-IBM

INTERVENTIONS:
Behavioral: M-IBM — In this paradigm, an ambiguous word or two-word phrase related to ASCC is followed by a sentence that resolves the word-sentence meaning as threatening or benign. For example, participants are presented with an ambiguous word or two-word phrase for 1 second. On half the trials the combination of the word/phrase and sentence creates a benign meaning (as in the previous example). On the other half of trials this combination creates an anxious-threat meaning Participants are required to judge the relatedness of the word/phrase and the sentence. Participants are given feedback during training such that judging the anxious-threat combinations to be "unrelated" and the benign combinations as being "related" would produce a "correct" response. In contrast, if participants produce an "incorrect" response they see "incorrect".
  Arms: M-IBM
Behavioral: Control-IBM — Placebo IBM where sentences are not related to anxious threat meaning of cue word.
  Arms: Control IBM

SUMMARY:
The Mobile-Interpretation Bias Modification clinical trial aims to examine the efficacy of a brief mobile phone delivered interpretation bias modification to reduce anxiety sensitivity cognitive concerns and suicidal ideation in National Guard Personnel. The investigators propose a randomized controlled trial testing the efficacy, acceptability, and usability of M-IBM with a sample of 114 National Guardsmen with current suicidal ideation and elevated anxiety sensitivity cognitive concerns. Participants will complete assessments, receive assistance on installing M- IBM on their phone, complete an M-IBM intervention session, and complete post-intervention assessments. Baseline measures of psychopathology, and usability/acceptability of M-IBM will be obtained during the initial session. In addition, 1-month, and 3-month follow-ups would be scheduled to examine changes in psychopathology. The investigators hypothesize that those randomized to M-IBM will experience reductions in anxiety sensitivity cognitive concerns, suicidal ideation. In addition participants will find M-IBM acceptable and easy to use.

ELIGIBILITY:
Inclusion Criteria:

* Elevated ASCC (>2) and include only Guard members who also have current SI (> 0) .
* Ownership of a smartphone

Exclusion Criteria:

* those determined by military or study personnel to be actively psychotic, manic, or imminently suicidal and in need of emergency services

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2019-12-15 (Actual); Primary Completion 2023-03-29 (Estimated); Study Completion 2023-03-29 (Estimated)

PRIMARY OUTCOMES:
Anxiety Sensitivity Index-3 Cognitive Concerns Subscale | 30 minutes
  Range 0 - 24, Higher Scores mean more pathology
Anxiety Sensitivity Index-3 Cognitive Concerns Subscale | 1 month post intervention
  Range 0 - 24, Higher Scores mean more pathology
Anxiety Sensitivity Index-3 Cognitive Concerns Subscale | 3 months post intervention
  Range 0 - 24, Higher Scores mean more pathology
The Self-Injurious Thoughts and Behaviors Interview | 1 month post intervention
The Self-Injurious Thoughts and Behaviors Interview | 3 months post intervention

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern Mississippi, Hattiesburg, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No